CLINICAL TRIAL: NCT04549740
Title: The Role of Salivary Alpha Amylase in Sepsis
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Other Study IDs: salivary amylase in sepsis
Record Dates: First submitted 2020-09-05; First posted 2020-09-16 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — venous sample will be withdrawn to estimate serum procalcitonin level. Saliva samples will be obtained to estimate salivary alpha amylase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: salivary alpha amylase level measurement — Saliva samples will be obtained to estimate salivary alpha amylase

SUMMARY:
Critical illness may be induced by different underlying life-threatening diseases, such as infection, sepsis, trauma, respiratory insufficiency or hypoxia and severe neurological status. The associated endocrine, nervous, metabolic and immunological changes are defined as acute stress syndrome. Salivary alpha-amylase is secreted from the salivary glands mainly in response to beta-adrenergic stimuli. Salivary alpha-amylase (sAA) has gained rapid popularity as a non-invasive marker of sympathetic nervous system (SNS) activity.

DETAILED DESCRIPTION:
Critical illness may be induced by different underlying life-threatening diseases, such as infection, sepsis, trauma, respiratory insufficiency or hypoxia and severe neurological status. The associated endocrine, nervous, metabolic and immunological changes are defined as acute stress syndrome.

Although sepsis is one of the oldest syndromes in medicine, it is a challenging healthcare problem even nowadays. In spite of the era of modern an¬tibiotics and intensive therapy sepsis is still one of the leading causes of morbidity and mortality.

Based on the novel results and advances of pathobiology, management and epidemiology of sepsis, the definitions of the syndrome have been changed recently. Sepsis-3 consensus de¬fines sepsis as a life-threatening organ dysfunc¬tion caused by a dysregulated host response to infection.

The diagnosis of sepsis is most often not easy especially in newborns or in patients whose im¬mune response is not adequate. Therefore, it is of most importance to introduce diagnostic biomarkers which can predict or verify systemic inflammation as early as possible. These tests should also be applicable for monitoring of the disease progression and efficacy of therapy as well.

Salivary alpha-amylase is secreted from the salivary glands mainly in response to beta-adrenergic stimuli.

Salivary alpha-amylase (sAA) has gained rapid popularity as a non-invasive marker of sympathetic nervous system (SNS) activity. sAA is a digestive enzyme that breaks down starch into glucose and maltose, and enzymatic activity (in Units/ml) is used as a proxy for sAA concentration.

The use of salivary alpha amylase as a marker of sympathetic activity seems justified. Salivary alpha amylase release from the salivary glands is under strong control of local sympathetic nerves. Its salivary concentration rapidly increases during acute stress, and its use as a marker of sympathetic activation is also validated by pharmacological studies.

ELIGIBILITY:
Inclusion Criteria:

* The newly diagnosed patients with sepsis according to Sepsis-3 consensus definition using SOFA score
* The newly diagnosed patients with septic shock according to Sepsis-3 consensus definition using SOFA score
* aged more than 18 years old.

Exclusion Criteria:

* Evidence of an immunocompromised as malignancy,
* received corticosteroids,
* recieved chemotherapy,
* recieved radiotherapy
* recieved cytotoxic drugs
* advanced hepatic disease
* renal disease
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The newly diagnosed patients with sepsis or septic shock according to Sepsis-3 consensus definition using SOFA score aged more than 18 years old.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
correlation of salivary amylase level and procalcitonin level in sepsis. | Through study completion average of 6 months
  correlation of salivary amylase level and procalcitonin level in the newly diagnosed patients with sepsis.

SECONDARY OUTCOMES:
correlation of salivary amylase level with mortality | during 28 follow up days of the patients
  correlation of salivary amylase level with mortality with follow up of the patients

CONTACTS AND LOCATIONS:
Locations (1):
- Tarek Abdel Hay, Tanta, El Gharbyia, Egypt